CLINICAL TRIAL: NCT06046846
Title: An Investigation of the Feasibility and Impact of a mHealth Prehabilitation Programme for Patients With Oesophago-gastric Cancer: The mPOC Study
Brief Title: Prehabilitation Via a Mobile Application in Oesophago-gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Alison Kelly, Principal Investigator, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 321301
Record Dates: First submitted 2023-07-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Oesophageal Cancer; Gastric Cancer; Prehabilitation; mHealth Application
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Single centred feasibility randomised controlled trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asensei app intervention group (Experimental): Participants randomised to the intervention group will be introduced to the mHealth prehabilitation programme delivered via a mobile app. Within this intervention group, participants will have access to a mHealth prehabilitation programme delivered and monitored via an app which will consist of a multimodal prehabilitation programme consisting of nutritional guidelines, improving well being and physical functioning prior to surgery.
  Interventions: Device: Asensei app
- Standard Pre-Operative Care group (No Intervention): The control group will receive standard pre-operative care within NHS Lothian for patients undergoing surgery for oesophago-gastric cancer which includes the enhanced recovery after surgery pathway. This pathway includes a pre-assessment, verbal advice only on prehabilitation interventions surrounding nutrition, well being and physical activity as well as a follow up post treatment.

INTERVENTIONS:
Device: Asensei app — The study will compare the delivery of a prehabilitation programme via a mHealth application against standard preoperative care for patients undergoing surgery for oesophago-gastric cancer
  Arms: Asensei app intervention group

SUMMARY:
The overall aim of this study is to assess the feasibility of a mHealth prehabilitation programme delivered via a mobile app for people with oesophago-gastric cancer by evaluating its user satisfaction and acceptance. The research question asks what is the feasibility of a mHealth prehabilitation programme delivered via a mobile app for patients with oesophago-gastric cancer?

The primary aim of this single centred feasibility randomised controlled trial (RCT) is to explore the recruitment, adherence, and compliance of taking part in a mHealth prehabilitation programme delivered for 6 weeks via a mobile app prior to oesophago-gastric surgery. This study will develop a prehabilitation programme to investigate the feasibility and impact of delivering prehabilitation via a mobile app to patients with a diagnosis of oesophago-gastric cancer before surgery.

DETAILED DESCRIPTION:
The study will test a six-week mHealth prehabilitation programme delivered via a modified mobile application called the asensei app. Asensei is a commercial company who have already successfully developed a digital platform known as the asensei app that delivers tailored training with individualised programmes and automated responsive feedback for the fitness industry via mobile applications. In summary, participants recruited to the study will require three visits to the hospital for measures to be taken. Outcome measurements will be taken at baseline (T0), prior to surgery (T1) and 30 days post surgery (T2). Outcome measures relating to feasibility, physical and nutritional functioning as well as quality of life will be collected at the above specified three time points (T0,1,2). There will also be weekly phone calls and one to one discussion after the six weeks of prehabilitation to explore how useful people have found the app and how easy and engaging it was to navigate. This study will gain valuable insight into the role mHealth applications could offer in preventing functional decline, improving quality of life and preventing secondary complications in patients with a diagnosis of cancer prior to surgery.

ELIGIBILITY:
Participants will need to fulfil the following eligibility criteria:

Inclusion Criteria:

* Diagnosis of oesophago-gastric cancer awaiting surgery,
* 18 years of age or over,
* Medically stable to participate in a prehabilitation programme with exercise intervention, English speaking,
* Access to an iPhone
* Able to provide informed consent.

Exclusion Criteria:

* Medically unstable,
* Diagnosis of metastatic cancer,
* Contraindications for physical activity,
* Presence of a pacemaker or other internal medical device,
* Uncontrolled blood pressure and or heart arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
To explore the recruitment of taking part in a mHealth prehabilitation programme delivered via the asensei app for 6-weeks prior to oesophago-gastric surgery. | Throughout the 6 weeks prior to surgery
  Recruitment will be measured by analysing the proportion of individuals who take up the offer of a mHealth prehabilitation programme delivered via the asensei app prior to surgical intervention.
To explore the adherence of taking part in a mHealth prehabilitation programme delivered via the asensei app for 6-weeks prior to oesophago-gastric surgery. | Throughout the 6 weeks prior to surgery
  Adherence with the mHealth prehabilitation will be calculated by analysing the percentage of participants who consistently engage with the asensei app and complete the prescribed prehabilitation programme.
To explore the compliance of taking part in a mHealth prehabilitation programme delivered via the asensei app for 6-weeks prior to oesophago-gastric surgery. | Throughout the 6 weeks prior to surgery
  Compliance will be measured by assessing the extent to which participants adhere to the recommended prehabilitation protocols as well as the study guidelines.
To investigate the fidelity in terms of user engagement of the asensei app to deliver a mHealth prehabilitation programme using the modified mobile application rating scale (mMARS). | The single point of assessment will be 30 days post surgery.
  Fidelity of the asensei app use will be measured using the modified mobile application rating scale (mMARS). This scale is a well-established framework for classifying and assessing the objective and subjective quality of apps. The scale assesses app quality which is rated on a 5-point scale from "1.Inadequate" to "5.Excellent". The modified mobile application rating scale typically ranges from 1 to 5, with 1 being the lowest rating and 5 being the highest. Higher scores generally indicate better user satisfaction and positive experiences with the mobile application. It suggests that users find the app to be more useful, user-friendly and enjoyable. Lower scores typically suggest dissatisfaction or negative experiences with the mobile application where users may find the app less useful, difficult to use or unenjoyable. Lower scores could also indicate issues with functionality, design or overall user experience.
To investigate the usability in terms of user satisfaction of the asensei app to deliver a mHealth prehabilitation programme. | The single point of assessment will be 30 days post surgery.
  Usability of the asensei app in terms of user satisfaction will be measured through semi structured interviews to collect participant feedback regarding the applications usability, perceived usefulness, and satisfaction. Higher and lower subjective ratings collated during the interview could represent different aspects of the app's performance and user experience. For example, a higher rating within interviews among participants may typically represent greater satisfaction with the mobile app with an increase likelihood to find the app user friendly, useful, and enjoyable to use. On the other hand, lower subjective feedback may typically signify dissatisfaction with the app.

SECONDARY OUTCOMES:
To investigate the incidence of treatment-emergent adverse events of using the mHealth prehabilitation programme delivered via the asensei app. | From 6 weeks prior to surgery to 30 days post surgery
  Any adverse effects of using the asensei app will be measured through participant monitoring via agreed weekly phone calls throughout the prehabilitation programme. These phone calls will collect data on any related treatment-emergent adverse events. Any reported events or concerns will be analysed systematically, and any events reported will be categorized according to severity, frequency, and the nature of the adverse effects.
To collect preliminary data on physical activity and assess for change using the Godin Leisure time Exercise questionnaire in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  Preliminary data on physical activity will subjectively measure physical activity using the self-administered Godin Leisure Time Exercise Questionnaire which is a validated self-reported physical activity measurement used in cancer care. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). The minimum and maximum values within the questionnaire used ranges from (0-119) where higher scores indicate higher level of leisure time exercise participation.
To collect preliminary data on aerobic capacity and assess for change using the 6 minute walk test (6MWT) in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The 6-minute walk test (6MWT) will assess the distance walked over 6 minutes as a sub-maximal test of aerobic capacity. This outcome measure will be used to determine changes in physical function levels and cardiorespiratory fitness. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). The minimum score is zero indicating that the participant was unable to walk any distance within the six minute time frame and the highest score is the distance walked by the participant in six minutes.
To collect preliminary data on a participants mobility and balance and assess for change using the timed up and go test (TUAG) in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The timed up and go test (TUAG) will assess a person's mobility and balance using the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). The lower the time score represents the shortest time taken to complete the task, indicating better mobility and functional ability. The higher the time score represents the longest time taken to complete the task suggesting potential mobility issues or functional limitations.
To collect preliminary data on a participants lower extremity strength and frailty and assess for change using the five times sit to stand test (5XSST) in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The Five times sit to stand test (5XSST) will assess lower extremity strength and frailty in patients with cancer. It is a simple test that evaluates the time taken to complete five repetitions of standing up from a seated position and sitting back down again. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). The lowest score is the shortest time taken to complete the task, indicating better lower body strength and mobility. The highest score is the longest time taken to complete the task, suggesting potential difficulties in lower body strength and functional mobility.
To collect preliminary data and assess for change on a participants anthropometry such as body composition in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  Anthropometry will be assessed as height, weight, and body composition. Body composition will be assessed and calculated using Body Mass Index in the standard manner as height and weight. These multiple measurements will be aggregated to arrive at one reported value (e.g., weight and height will be combined to report BMI in kg/m) This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2).
To collect preliminary data and assess for change on a participants handgrip strength using the hand dynamometer in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The handgrip test will be assessed and measured using a hand dynamometer to assess for grip strength. Handgrip strength can be used in cancer patients to evaluate nutritional risk and the need for nutritional intervention. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). It measures the maximum force a person can generate while squeezing a handgrip dynamometer. The score is typically measured in kilograms and indicates the strength of the participants hand muscles. The lowest score is the weakest grip strength measurement achieved by the participant and the highest score is the strongest grip strength measurement obtained during the test.
To collect preliminary data and assess for change on a participants risk of malnutrition by using PG-SGA questionnaire in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The Patient Generated Subjective Global Assessment questionnaire (PG-SGA) will be used as an assessment tool to identify those most at risk of malnutrition. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). It does not have a specific numerical score range like some other tests. Instead it involves a series of questions and assessments that are used to evaluate a participants weight changes, dietary intake, symptoms and functional capacity. The results are typically categorised into different levels of malnutrition of nutritional risk, ranging from well nourished to severely malnourished.
To collect preliminary data and assess for change on a participants wellbeing by using the patient health questionnaire (PHQ-9) in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The patient health questionnaire (PHQ-9) will be used as an assessment tool to identify those participants in need of further support out with the universal programme provided by the asensei app. This will be assessed for change at three different time points: at baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). The PHQ-9 is a self assessment tool used to screen and assess the severity of depression. It consists of nine questions that measure the frequency of various depressive symptoms over the past two weeks. The PHQ-9 scores range from 0-27, with higher scores indicating greater severity of depressive symptoms and the lowest score is 0 indicating the absence of depressive symptoms.
To collect preliminary data and assess for change on a participants quality of life by using the EORTC QLQ-OG25 questionnaire in order to inform the sample size for a fully powered RCT as part of the feasibility study. | From 6 weeks prior to surgery to 30 days post surgery
  The EORTC QLQ-OG25 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire- Oesophagogastric Module 25) is a validated screening tool used in the quality-of-life metric pilots for patients with oesophageal-gastric cancer to be assessed for change at three different time points: baseline (T0), pre surgery (T1) and 30 days post-surgery (T2). The scoring for the EORTC QLQ-OG25 questionnaire is not a simple numerical range. It involves transforming raw scores into a scale of 0 to 100, where higher scores represent better functioning or higher levels of symptomatology, depending on the question. For example, higher scores on functional scales indicate better function and well-being, while higher scores on symptom scales indicate more severe symptoms. The scores are then interpreted in relation to the patient's condition and the context of their cancer diagnosis and treatment.

OTHER OUTCOMES:
Semi structured interviews | 30 days post surgery
  To collect insights into participants views on positive and negative experiences or impacts and thoughts on the asensei app and prehabilitation programme participation. Positive and negative experiences within a qualitative interview may indicate higher or lower ratings associated with the mobile app. For example, positive feedback may indicate that participants are more likely to recommend the app to others, which is a valuable indicator of user satisfaction and potential for growth. Negative feedback may reflect user frustration with the app's performance or limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Kelly, MRes, Principal Investigator — Queen Margaret University; Dr Gillian Baer, PhD, Study Director — Queen Margaret University

IPD SHARING:
Plan to Share IPD: Yes
Overall study outcomes will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available as part of a publication which is expected to be 31/12/2025 at the latest.
Access Criteria: The access criteria in which the Individual Participant Data (IPD) and any additional supporting information will be shared will become available after publication when summary data are published and otherwise made available. The journal with whom this will be made available is currently undecided.

REFERENCES:
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Zelenko O, Tjondronegoro D, Mani M. Mobile app rating scale: a new tool for assessing the quality of health mobile apps. JMIR Mhealth Uhealth. 2015 Mar 11;3(1):e27. doi: 10.2196/mhealth.3422. PMID 25760773
- [Background] Crans GG, Shuster JJ. How conservative is Fisher's exact test? A quantitative evaluation of the two-sample comparative binomial trial. Stat Med. 2008 Aug 15;27(18):3598-611. doi: 10.1002/sim.3221. PMID 18338319